CLINICAL TRIAL: NCT05567991
Title: Improving Stress Management, Anxiety, and Mental Well-being in Medical Students Through an Online Mindfulness-Based Intervention: a Randomized Study
Brief Title: Studying the Effect of a Mindfulness-based Intervention on Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Teresa Fazia, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1Med_a
Record Dates: First submitted 2022-09-14; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Mental Well-being
Keywords: mindfulness; well-being; medical students; distress; resilience; emotion regulation
MeSH Terms: conditions — Psychological Well-Being; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The individuals assigned to the treatment group attend the training sessions and were asked to complete all the questionnaires at both time points
  Interventions: Behavioral: Comprehensive Mindulness-Based Intervention (C-MBI)
- Passive Control Group (No Intervention): The individuals assigned to the passive control group did not attend any training session and were only asked to complete the same questionnaires as the treatment group at both time points. Participants in the control group were asked not to practice meditation during the period of the study for an unbiased comparison with the intervention group.

INTERVENTIONS:
Behavioral: Comprehensive Mindulness-Based Intervention (C-MBI) — C-MBI, was administer online via Zoom and included: 10 Integral Meditation classes lasting approximately 35 minutes each, given twice a week (Monday and Wednesday); 10 minutes of yoga exercises focused on breathing and posture before each IM class; and dietary advice. Regarding this latter, the participants received via email a document which entailed non-mandatory dietary suggestions to promote healthy nutrition, sleep and stress-relief. An online lecture held by the nutritionist with a question-and-answer format was also organized. The degree to which to follow this advice was left to the discretion of each participant. The core of our intervention was represented by the IM training, that is a MBI intervention, that simultaneously uses breathing, focusing attention, releasing of physical tensions, thoughts and feeling sensations through internal senses and imagery, allowing a quick relaxation and more deeply a physical, energetic, and spiritual well-being.
  Arms: Treatment group

SUMMARY:
In the scientific literature, the responsibilities and pressures of medical school and residency are widely known for putting a strain on medical student's personal wellbeing, leading to high rates of anxiety, depression, burnout, and emotional discomfort. In this study investigators aim at evaluating the hypotheses on the effectiveness of a comprehensive Mindfulness-Based Intervention (MBI) in reducing this load. The intervention comprised 12 Integral Meditation (IM) classes, advice on health dietary behavior and brief yoga session. The effect of the intervention on medical students from Italian universities will be evaluated by performing a randomized trial through the analysis of nine questionnaires used for measuring the psychological outcomes of interest.

DETAILED DESCRIPTION:
In the scientific literature, the responsibilities and pressures of medical school and residency are widely known for putting a strain on medical student's personal wellbeing, leading to high rates of anxiety, depression, burnout, and emotional discomfort. Academic pressure, financial concerns, workload, sleep deprivation, drugs abuse, exposure to patients' suffering and fatalities are among the numerous causes linked to such a decrease in mental well-being in medical studies setting. The so-called hidden curriculum is also a factor considered in medical education. It is based on implicit teaching that includes moral and ethical values among medical education. When this teaching goes in a negative direction such as cynicism towards patients, future career, or competition with colleagues, can become one of the causes that influences medical students in terms of psychological distress and burnout. Additionally, psychological distress among students has been claimed to have a negative impact on their academic performance, and on the increased thought of dropping out medical school. This also leads to academic dishonesty, which includes problems such as plagiarism, cheating, pseudoscience and falsification, and to alcohol and substance addiction. Medical students suffering from psychological distress have a more generally lack of empathy.

To make matters worse, the recent Covid-19 pandemic has placed an additional burden on students around the world Aware of this situation, medical students are using different coping strategies to reduce distress. While taking drugs and substances such as tranquilizers, have negative or side effects, taking social support and physical activity have positive effects only. Mindfulness-Based Interventions (MBI) is an effective complement to these strategies.

Mindfulness is a state of pre-reflexive consciousness that can be put in contrast with other modalities in which the person is constantly engaged in overthinking, obsessing about the past, fantasizing and worrying about the future or engaged in compulsive or automatic behavior without acknowledging it. The benefits of such a state of being is well-known in literature, so that MBIs are getting popular in medical education, to such an extent that many medical schools around the world are beginning to acknowledge mindfulness as a helpful practice for their students, residents, and staff with the goal of also increase patient care quality.

Hence to develop and apply easily accessible and low-cost strategies to diminish the levels of stress of medical students is crucial for their academic performance and professional development.

The aim of the present study was to assess the efficacy of a comprehensive MBI, entirely administered online, consisting of a mindfulness-based practice, called Integral Meditation (IM), dietary advice, and brief yoga sessions, in two cohorts of Italian medical students randomized to intervention or control group. The primary hypothesis is that participants in the intervention group would report a decrease of perceived stress and state anxiety and an increase of mental well-being. The secondary hypothesis investigators tested was that participants in the intervention group would report higher scores on different measures of positive affect, resilience, and emotion regulation and attentional control. The investigated outcomes were measured using nine self-report questionnaires administered online to both groups before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must have digital advice and an Internet connection to complete the assessment and to attend the classes
* Must understand Italian language

Exclusion Criteria:

* Severe anxiety or depression
* Severe mental illness (e.g., hypomania or psychotic episode)
* Any other serious mental or physical health problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2021-01-23 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
change in perceived stress | Assessed at baseline (to) and after the intervention (12 weeks)
  Perceived stress outcome will be measured through the Perceived Stress Score (PSS) questionnaire. PSS can range from 0 to 40 with higher scores indicating higher perceived stress. The scores obtained from the questionnaire is a measure of the psychological investigated outcome.
Change in state anxiety | Assessed at baseline (to) and after the intervention (12 weeks)
  The state anxiety outcome will be measured through the State Anxiety Inventory (STAI-X1) questionnaire. Score ranges from 0-63 with higher scores indicating higher state anxiety levels. The scores obtained from the questionnaire is a measure of the psychological investigated outcome.
Change in mental well-being | Assessed at baseline (to) and after the intervention (12 weeks)
  The well-being outcome will be measured through the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) questionnaire. Higher scores indicate mental well-being. PSS can range from 14 to 70 with higher scores indicating higher well-being. The scores obtained from the questionnaire is a measure of the psychological investigated outcome.

SECONDARY OUTCOMES:
Change in positive affect | Assessed at baseline (t0) and after the intervention (12 weeks)
  Positive affect outcome through Positive and Negative Affect Schedule (PANAS) measuring both Positive affect (PA) and Negative affect (NA). Scores range 10-50 for both. Higher PA score indicates more positive affect, while lower NA score less negative affect.
Change in resilience | Assessed at baseline (t0) and after the intervention (12 weeks)
  Resilience through the Resilience Scale (RS-14) that ranges 14-98, higher scores indicate a higher level of resilience.
Change in mind-wondering | Assessed at baseline (t0) and after the intervention (12 weeks)
  Mind-wondering outcome through Mind Wandering Spontaneous (MW-S) that ranges 4-28, higher score indicating a higher tendency of mind wandering in daily life.
Change in emotion regulation | Assessed at baseline (t0) and after the intervention (12 weeks)
  Emotion regulation outcome through Difficulties in Emotion Regulation Scale (DERS). Scores range 33-165, higher score indicates higher difficulties in emotion regulation
Change in attentional control | Assessed at baseline (t0) and after the intervention (12 weeks)
  Attention control outcome through Attention Control (AC-S and AC-W) Scales that range 4-20 and 4-40, higher score indicating higher attentional distraction and difficulties in attentional shifting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavia, Pavia, Italy